CLINICAL TRIAL: NCT05327751
Title: Possible Protective Effect of Celecoxib Against Capecitabine Induced Hand and Foot Syndrome in Patients With Colorectal Cancer
Acronym: HFS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Kettana, clinical pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 42022
Record Dates: First submitted 2022-04-01; First posted 2022-04-14 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Hand and Foot Syndrome; Erythrodysesthesia Syndrome; HFS; Colorectal Cancer
Keywords: capecitapine induced hand and foot syndrome; Hand and Foot Syndrome; Erythrodysesthesia Syndrome; HFS; capecitabine based chemotherapy; Colorectal Cancer
MeSH Terms: conditions — Hand-Foot Syndrome; Colorectal Neoplasms | interventions — Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celecoxib arm (Active Comparator): This arm will include 22 patients who will receive 6 cycles of capecitabine-based chemotherapy (cycle is every 3 weeks) in addition to 200 mg of oral celecoxib twice daily for 14 days of the 3-week cycle. The study duration will be the duration of the 6 cycles.
  Interventions: Drug: Celecoxib 200mg; Drug: Capecitabine-based chemotherapy
- Control arm (Placebo Comparator): This arm will include 22 patients who will receive 6 cycles of capecitabine-based chemotherapy (cycle is every 3 weeks).
  Interventions: Drug: Capecitabine-based chemotherapy

INTERVENTIONS:
Drug: Celecoxib 200mg — 200 mg of oral celecoxib twice daily for 14 days of the 3-week cycle.
  Arms: Celecoxib arm
Drug: Capecitabine-based chemotherapy — Capecitabine-based chemotherapy

SUMMARY:
Colorectal cancer (CRC) is the third most common cancer and the second leading cause of malignancy-related mortality. Capecitabine has been approved for the treatment of colorectal cancer as first-line therapy. About 50%-68% of patients who take capecitabine develop Hand-foot syndrome. Hand-foot syndrome (HFS) is the most common adverse event of capecitabine-based chemotherapy. Initial symptoms of HFS are dysesthesia, tingling in the palms, fingers, and soles of the feet, and erythema, which may progress to an extremely painful and debilitating condition without prompt management. These symptoms can potentially lead to a worsened quality of life in patients taking capecitabine-based chemotherapy. Moreover, the adverse reaction necessitates dose-reduction or withdrawal of the chemotherapeutic agent. The mechanisms of HFS are still unknown, and there are limited data available on how to prevent them or manage them. However, different hypotheses of capecitabine-induced HFS pathogenesis have been suggested. One of the hypotheses stated that HFS is a kind of inflammation mediated by cyclooxygenase's (COX-2) over expression in palm and feet by capecitabine and its metabolites causing elevation of inflammatory markers as tumor necrosis factor alpha (TNF-α). COX-2 enzyme plays a main role in inflammation and pain. Therefore, celecoxib which is selective (COX-2) inhibitor may have a key role in the HFS treatment plan. A retrospective study and two prospective studies showed that combining capecitabine with celecoxib, a selective COX-2 inhibitor, can significantly reduce capecitabine-related HFS in colorectal cancer patients. Those studies were dependent on HFS grading only without measuring any markers. So, in our study we assess possible protective effect of celecoxib against capecitabine induced HFS and measure inflammatory marker as tumor necrosis factor alpha (TNF-α), oxidative stress marker as Malondialdehyde (MDA), and cyclooxygenase-2 (COX-2) enzyme to show whether capecitabine induced HFS is caused by COX-2 mediated inflammation or not.

ELIGIBILITY:
Inclusion criteria:

* Age: 18-65 years old.
* Gender: Male and female.
* Newly diagnosed colorectal cancer patients who are scheduled to receive capecitabine-based chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Patients with adequate renal function (Sr. creatinine < 1.2 mg/dl or eGFR ≥ 90 ml/min).
* Patients with adequate hepatic function (Sr. bilirubin < 1.2 mg/dl).

Exclusion criteria:

* Pregnant and lactating females.
* Patients with cardiovascular disease (congestive heart failure, cardiac arrhythmia, or coronary artery disease, …. etc.).
* History of H-Pylori infection.
* Patients with a known hypersensitivity to any of the used drugs.
* Patients with any contraindication to any of the used drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The change in HFS grading. | After each cycle (each cycle is 21 days).
  The change in hand and foot syndrome (HFS) grading according to common terminology criteria of adverse events (CTCAE) version 5.0.
The change in HFS-specific QOL questionnaire (HFS-14). | After each cycle (each cycle is 21 days).
  Assessment of patients' quality of life using HFS-specific QOL questionnaire (HFS-14) based on patients' symptoms.

SECONDARY OUTCOMES:
The change in serum levels of cyclooxygenase-2 (COX-2) enzyme. | At basline and after the sixth cycle (each cycle is 21 days).
  The change in serum levels of cyclooxygenase-2 (COX-2) enzyme.
The change in serum levels of tumor necrosis factor alpha (TNF-α). | At basline and after the sixth cycle (each cycle is 21 days).
  The change in serum levels of tumor necrosis factor alpha (TNF-α) as a inflammatory marker.
The change in serum levels of malondialdehyde (MDA). | At basline and after the sixth cycle (each cycle is 21 days).
  The change in serum levels of malondialdehyde (MDA) as oxidative stress marker.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Pharmacy-Tanta University, Tanta, Egypt